CLINICAL TRIAL: NCT06542523
Title: Observational Study Regarding the Necessity of Inclusion of Foot Arch State Together With the Angiosome Theory Within the Wound, Ischemia and Foot Infection Classification (WIfI) to Enhance the Predictability of Wound Healing and Decision Making
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: AinShamsUnivascular
Record Dates: First submitted 2024-06-26; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-02

CONDITIONS: Chronic Limb-Threatening Ischemia; Diabetic Foot; Vascular Diseases
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetic Foot; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (15):
- WIFI stage 1 with type 1 foot arch
- WIFI stage 2 with type 1 foot arch
- WIFI stage 3 with type 1 foot arch
- WIFI stage 1 with type 2a foot arch
- WIFI stage 2 with type 2a foot arch
- WIFI stage 3 with type 2a foot arch
- WIFI stage 1 with type 2b foot arch
- WIFI stage 2 with type 2b foot arch
- WIFI stage 3 with type 2b foot arch
- WIFI stage 1 with type 3a foot arch
- WIFI stage 2 with type 3a foot arch
- WIFI stage 3 with type 3a foot arch
- WIFI stage 1 with type 3b foot arch
- WIFI stage 2 with type 3b foot arch
- WIFI stage 3 with type 3b foot arch

SUMMARY:
This study aims to assess the complete healing or healing progress of foot ulcer within 1 year Where the patients will be classified according to foot arch state together with the angiosome theory and the WIFI clinical stage to reflect the the necessity of inclusion of foot arch state together with the angiosome theory within the WIFI classification to enhance the predictability of wound healing and decision making

DETAILED DESCRIPTION:
Patients will be classified according to their WIFi stages into 3 groups and each group will be furtherly classified according to the patient's angiography of foot arch (whether by CT angiography or direct angiography) into:

Type 1: patent foot arch Type 2: partially occluded foot arch which is divided into whether Type 2a: patent dorsal tributary of foot arch Type 2b: patent lateral tributary of foot arch Type 3: totally occluded foot arch is divided into whether. Type 3a: totally occluded foot arch with anterior tibial artery inflow. Type 3b: totally occluded foot arch with posterior tibial artery inflow.

During follow-up assessments, wound is classified to be within: anterior tibial artery, posterior tibial artery or both territories.

Wound healing states are often classified based on the progression of the healing process into each of the following categories such as:

1. Complete Healing: Wound closure with the restoration of tissue integrity and absence of signs of infection.
2. Partial Healing: Significant improvement but not complete closure; may involve reduction in wound size and improved tissue viability.
3. Worsening: Increase in wound size or signs of infection which may necessitates performing major amputation.

ELIGIBILITY:
Inclusion Criteria:

* diabetic foot in the form of gangrene, or a lower limb ulceration >2 weeks duration.

Exclusion Criteria:

1. Age below 18 years old.
2. Critically ill patients
3. Patients with acute ischemia
4. patients with pure venous ulcer
5. patients with ulcer due to rheumatological disease
6. The patient has known sensitivity to heparin.
7. The patient has comorbid conditions that may limit their ability to comply with the follow-up requirements
8. The patient has an untreatable allergy to radiographic contrast material.
9. Patient refusing consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients walking in or referred to the out-patient clinic at Ain Shams University Specialized Hospitals or El-Demerdash University Hospitals with symptoms of diabetic foot ulcer or gangrene.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Complete Healing | 2,4,6 months
  Wound closure with the restoration of tissue integrity and absence of signs of infection.
Partial Healing: | 2,4,6 months
  significant improvement but not complete closure; may involve change in wound size and improved tissue viability.
Worsening | 2,4,6 months
  change in wound size or signs of infection which may necessitates performing major amputation. .

SECONDARY OUTCOMES:
Occurrence of Complication | within 30 days of the procedure
  Rates of procedure- and device-related adverse events during revasularization

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt